CLINICAL TRIAL: NCT03597035
Title: Mineralocorticoid Receptor Antagonism Clinical Evaluation in Atherosclerosis Add-On
Acronym: MAGMAAddOn
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study could not enroll patients owing to the inclusion exclusion criteria
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Relypsa, Inc. (Industry)
Responsible Party: Principal Investigator, Sanjay Rajagopalan, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-17-16
Record Dates: First submitted 2018-03-05; First posted 2018-07-24 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Type2 Diabetes; Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — Spironolactone; patiromer

STUDY DESIGN:
Intervention Model Description: An open label proof-of-concept clinical trial in 50 patients with Type II diabetes evaluating the effects of MRA + Patiromer on LV mass and plaque regression over 12 months of treatment by magnetic resonance imaging (MRI).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patiromer Add-On (Experimental): Single arm experimental study in 50 diabetic patients with chronic kidney disease and hyperkalemia.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — The study participants will receive concomitant treatment with Veltassa 8.4 grams per day and Spironolactone 25 mg per day or maximum tolerated dose. If dictated by the potassium level, Veltassa can be increased to 16.8 grams per day.
  Other Names: Veltassa

SUMMARY:
Patiromer add-on to a mineralocorticoid receptor antagonist (MRA) in patients with Type 2 diabetes mellitus and chronic kidney disease (CKD) will reduce blood pressure and left ventricular (LV) mass to a greater extent compared to patients with MRA alone and favorably affect key secondary hemodynamic and inflammatory variables including atherosclerosis progression.

Atherosclerosis is the leading cause of morbidity and mortality in Type II diabetes. A cell type called the monocyte/macrophage is critical to development and complications of atherosclerosis.

This project will evaluate the effectiveness of a medication called Spironolactone in addition to Patiromer in preventing atherosclerosis in Type II diabetes through its effects on cells such as the monocyte. Spironolactone has been demonstrated to be effective for the treatment of patients after a heart attack and stroke. The investigators will evaluate the impact of Spironolactone in combination with Patiromer in reducing atherosclerosis plaque and additionally evaluate its potential in changing inflammation.

The investigators envision that a strategy of simultaneously probing effect of a drug combined with analysis of mechanisms of action and predictive response will likely provide key information with which to design hard event (heart attack, stroke etc.) based trials.

DETAILED DESCRIPTION:
There is substantial interest in preventing cardiovascular (CV) and renal disease progression in the Type 2 diabetic. Activation of the renin angiotensin aldosterone axis (RAS) and the mineralocorticoid receptor (MR) results in pro-inflammatory effects. Further the phenomenon of aldosterone escape provides a rationale for MR antagonism in addition to an ACEI/ARB agent. Agents that target the renin-angiotensin aldosterone system (RAAS) cascade have shown benefit in Type 2 Diabetics although combined RAS blockade such as using ACEI+ARB or ACEI/ARB+Renin inhibition have met with failure primarily owing to adverse effects such as hypotension and renal failure/hyperkalemia requiring dialysis. It has been speculated that dual RAS blockade or use of ACEI/ARB in conjunction with MRA may potentially be beneficial if one controls hyperkalemia and/or avoid excess hypotension. As a foundation for this current proposal, the investigators have demonstrated an important role for RAAS and MR antagonism in reducing atherosclerosis and inflammation in experimental animal models and limited studies in humans. The investigators are currently testing the efficacy of Spironolactone in reducing atherosclerosis on top of ACEI/ARB in high-risk patients with type 2 diabetes (T2DM) with concomitant CKD as part of a Randomized Double-blind controlled clinical trial. Given the fact that as much as 20-40% of a diabetic patient population with CKD may have problems of hyperkalemia on spironolactone, particularly those already on angiotensin converting enzyme inhibitor (ACEI)/ARB therapy, that would preclude their participation in this trial, the investigators would like to propose an open label supplemental arm to where patients who are ineligible for participation owing to baseline hyperkalemia or hyperkalemia on the dose escalation phase will be eligible to participate in the PRIMARY-Add on trial. The addition of Patiromer will enable introduction of MRA therapy at therapeutic doses and avoidance of hyperkalemia. The investigators thus propose a prospective open label trial with blinded assessment of end-points (PROBE) study which test the relative safety and efficacy of Patiromer on top of Spironolactone in T2DM on LV mass regression and occurrence of hypokalemia (Co-Primary End-points) as well as its effect on 24-hour ambulatory blood pressure (ABP) at 6 weeks, central aortic blood pressure at 6 weeks, atherosclerosis progression at 12 months and measures of monocyte inflammatory potential. If successful, the studies outlined in this proposal will extend the utility of Patiromer in high-risk diabetics at risk for future CV events and provide new information.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients >= 45 years and able to provide informed consent (females must be either post-menopausal for one year, surgically sterile, or using effective contraception. Oral contraceptives are disallowed.)
2. Patients with type II diabetes with HbA1c ≤ 9.0 on stable anti-glycemic regimen that may include oral and/or injectable therapy (GLP-1/Insulin etc.). Changes in dose of glycemic regimen is allowed during the course of the trial if felt to be clinically appropriate.
3. Glomerular filtration rate (GFR) <90 and evidence of proteinuria (Urine Albumin/Creatinine Ratio of >30 mg/g or equivalent) in a urine specimen within 12 months OR GFR <60 mg/g regardless of proteinuria
4. Patients must be on angiotensin-converting-enzyme inhibitor (ACE) and/or angiotensin-resistance-blocker (ARB) therapy with no planned dose adjustments.
5. Hyperkalemia defined as serum K+≥ 5.1 meq/L at visit 0 (screening).

Exclusion Criteria

1. Uncontrolled hypertension (Systolic Blood Pressure (SBP)>160 and/or Diastolic Blood Pressure (DBP)>95 mmHg at visit 0 (screening) and SBP >145 mm Hg at visit 2).
2. GFR (MDRD) of <20 at visit 0 (screening)
3. Hyperkalemia defined as serum K+ <5.1 meq/L at visit 0 (screening).
4. LDL cholesterol >150 mg/dL
5. Plasma triglycerides > 400 mg/dl
6. Contraindications to MRI (metallic implants, severe claustrophobia).
7. Acute coronary syndrome, Transient ischemic attack, cardiovascular accident (CVA) or critical limb ischemia during the last 6 months or coronary/peripheral revascularization within the last 3 months.
8. Evidence of a secondary form of hypertension.
9. Initiation of new therapy with statins, ACE/ARB, antioxidants, calcium channel blockers (CCBs), diuretics, β blockers.
10. Type I diabetes mellitus
11. Known contraindication, including history of allergy to Spironolactone or Patiromer
12. Any surgical or medical condition which might alter pharmacokinetics of drug (e.g. renal transplant, liver failure, liver transplant)
13. Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia.
14. Significant hyponatremia defined as Na <130 meq/L.
15. History of prior malignancy including leukemia and lymphoma (but not basal cell skin cancer, cured squamous cell cancer and cured prostate cancer).
16. History of any severe, life-threatening disease.
17. Any surgical or medical conditions which place the patient at higher risk derived from his/her participation into the study, or likely to prevent patient from complying with requirements.
18. History of drug abuse within the last 2 years, noncompliance and unwillingness/inability to consent.
19. Pregnant women and nursing mothers
20. Class III or IV Congestive Heart Failure
21. Primary Hyperaldosteronism

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Rajagopalan, MBBS, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single arm experimental study in 50 diabetic patients with chronic kidney disease and hyperkalemia.
  Spironolactone: The study participants will receive concomitant treatment with Veltassa 8.4 grams per day and Spironolactone 25 mg per day or maximum tolerated dose. If dictated by the potassium level
Period: Overall Study
Arm/Group | Patiromer Add-On
Started | 8
Completed | 4
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Patiromer Add-On
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 66 [56 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Mass
Description: Change in left ventricular mass from baseline to 12 months.
Time Frame: Time 0: study baseline, beginning of treatment. Time 1: 12 months follow-up, end of treatment.
Population: Data not collected
Groups:
- Spironolactone: Participants are to receive up to 25mg of spironolactone and 16.8g/d of patiromer.
- Placebo: Participants are to receive up to 25mg of placebo and 16.8g/d of patiromer.
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Patiromer Add-On
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03597035/Prot_SAP_000.pdf